CLINICAL TRIAL: NCT06661538
Title: Addressing Food Insecurity in the Health Care Setting to Promote Health Equity
Brief Title: Implementing Food Referrals for Equity and Sustained Health
Acronym: I-FRESH
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Rady Children's Hospital, San Diego (Other)
Responsible Party: Principal Investigator, Kay Rhee, Professor, University of California, San Diego
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: IRB # 810869; R01DK140573 (NIH)
Record Dates: First submitted 2024-10-17; First posted 2024-10-28 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Food Insecurity
Keywords: Food Insecurity; Social Care; Screening; Type 2 Diabetes Mellitus; Cardiovascular Disease; Child Health; Nutrition; Fruit and Vegetables; Care Navigation; Metabolic Dysfunction-Associated Steatotic Liver Disease; NAFLD; Nutrition Support Programs
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Intervention Model Description: This is a pilot type 2 hybrid effectiveness-implementation trial of the I-FRESH program using the Roll-out Implementation and Optimization (ROIO) design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Clinic 1: Type 2 Diabetes Clinic (Experimental): Families with children who attend the Type 2 Diabetes Clinic and indicate that they are experiencing food insecurity on the 2-item screener will be eligible for participation in this group.
  Interventions: Behavioral: Food Security Screening & Referral Program
- Clinic 2: Obesity Clinic (Experimental): Families with children who attend the Obesity Clinic in Endocrinology and indicate that they are experiencing food insecurity on the 2-item screener will be eligible for participation in this group.
  Interventions: Behavioral: Food Security Screening & Referral Program
- Clinic 3: Preventive Cardiology Clinic (Experimental): Families with children who attend the Preventive Cardiology Clinic for hypertension and/or high cholesterol and indicate that they are experiencing food insecurity on the 2-item screener will be eligible for participation in this group.
  Interventions: Behavioral: Food Security Screening & Referral Program
- Clinic 4: Gastroenterology Clinic (Experimental): Families with children who attend the Gastroenterology Clinic for malnutrition or MASLD and indicate that they are experiencing food insecurity on the 2-item screener will be eligible for participation in this group.
  Interventions: Behavioral: Food Security Screening & Referral Program

INTERVENTIONS:
Behavioral: Food Security Screening & Referral Program — The I-FRESH (Implementing Food Referrals for Equity and Sustained Health) program is the food security nutrition support program that involves some combination and form of: 1) screening and identification of families experiencing food insecurity; 2) discussions with families to determine readiness to engage with nutrition support programs and other community resources; 3) referrals and support to engage with a program; and 4) conducting follow-up assessments to determine fit of program, track utilization, and assess need for additional referrals. The exact implementation and workflow for this program will be optimized for each clinic.

SUMMARY:
Food insecurity (FI) disproportionately affects those who have been historically marginalized and significantly contributes to poor health outcomes. In children, FI is associated with lower psychosocial functioning and academic achievement. It also contributes to the development of adverse health outcomes such as obesity, type 2 diabetes mellitus (T2DM), cardiovascular disease (CVD), and Metabolic Dysfunction-Associated Steatotic Liver Disease (MASLD). Improving the diet quality of children (e.g., decreasing fat intake, increasing fruits and vegetables (FV) and fiber intake) has been associated with lower fasting serum glucose, insulin, LDL cholesterol, non-HDL cholesterol, and reduced risk of CVD later in life. Increasing awareness and access to programs that promote food equity by providing affordable healthy produce is a promising way to improve health outcomes and empower patients and communities to achieve better health and well-being. The goal of this proposal is to refine and optimize implementation strategies that connect families to community-based food security nutrition support programs through health care systems or medical clinics. The investigators will develop a multi-disciplinary, cross-sector collaboration to optimize current processes and workflows that integrate food security nutrition support programs into the healthcare system. The investigators will also work to develop a closed-loop communication system between the healthcare and healthy food access systems to support greater patient autonomy and self-efficacy to obtain, prepare, and consume healthy foods.

DETAILED DESCRIPTION:
The investigators will conduct a pilot type 2 hybrid effectiveness-implementation trial of the I-FRESH (Implementing Food Referrals for Equity and Sustained Health) program using a Roll-Out Implementation Optimization (ROIO) design among families with children with nutrition-related illnesses who receive Medicaid or Supplemental Nutrition Assistance Program (SNAP) benefits. The I-FRESH program, the food security nutrition support program, will be refined prior to the first clinic roll-out based on input from several hospital, clinical, and community stakeholders. The program will involve 4 main components: screening and identification of families experiencing food insecurity (FI); social worker/care navigator-led discussions with families to determine need and readiness to receive support; referrals and assistance to engage with these programs; and follow-up assessments to determine fit, track utilization, and determine need for additional referrals. With each roll-out into a new clinic, modified implementation procedures and work-flows will be evaluated using implementation and effectiveness outcomes.

ELIGIBILITY:
Inclusion Criteria:

* child attending Type 1 or Type 2 Diabetes clinics, Cardiology clinic, MASLD clinic, general GI clinic at RCHSD
* child age between 5-18 years old
* parent or caregiver who indicates that they are experiencing food insecurity and receives Medicaid or SNAP benefits
* family not moving out of the San Diego area within the time frame of the study

Limited exclusion criteria will be applied in order to examine the impact of this program on a heterogenous group of people and increase generalizability. Of note, all genders and races/ethnicities will be allowed to participate.

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2027-06-15 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Intervention Measure (FIM) | 12 months
  4-item measure that assesses feasibility of implementing the program in that setting; score range (4-20) with higher scores referring to greater feasibility
Acceptability of Intervention Measure (AIM) | 12 months
  4-item measure assessing the acceptability of the program by program staff and participants; score range (4-20) with higher scores referring to greater acceptability
Implementation Fidelity | 12 months
  Percent of families with food insecurity that were called, percent of families that were referred to a program or provided with resources, percent of families that received follow-up phone calls, percent of families that needed additional resources/referrals
Adoption | 12 months
  Percent of clinical settings approached that participate; characteristics of settings participating compared to non participating clinical settings
Reach | 12 months
  Percent of families attending clinic that completed the food insecurity screener, number of families experiencing food insecurity in that clinic, percent of families that wanted and did not want referrals to a nutrition support program

SECONDARY OUTCOMES:
Change in Food Security levels over a 12 month period | 12 months
  U.S. Household Food Security Survey Module: Six-Item Short Form; Score range of 0-6, with higher scores indicating greater food insecurity
Change in Weight Status over 12 months | 12 months
  Weight status may be measured by BMI percentile for age and sex, %BMIp95, %BMIp50, or BMI z-score
Change in Blood Pressure over 12 months | 12 months
  Change in systolic and diastolic blood pressures
Change in non-fasting and fasting Lipid levels over 12 months | 12 months
  Change in total cholesterol, non-HDL cholesterol, HDL cholesterol, triglycerides, and LDL cholesterol
Change in HbA1c over 12 months | 12 months
  change in HbA1c levels over a 12 month period
Change in Liver Function Tests over 12 months | 12 months
  change in AST and ALT over a 12 month period
Change in Quality of Life measure over 12 months | 12 months
  Parent reported Quality of Life as measured by the Pediatric Quality of Life Inventory (PedsQL); Score range of 0 to 100, with higher scores indicating a higher quality of life

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - UC San Diego, La Jolla, California
  - Rady Children's Hospital San Diego, San Diego, California

IPD SHARING:
Plan to Share IPD: Yes
We will make a complete description of our final study protocol available at the end of the study. We will provide details regarding our study population (inclusion and exclusion criteria as well as demographic information) and describe our strategy for engaging patients, clinicians, and other stakeholders in the design and implementation of this program. We will make available our workflows and specific measurement tools. The program protocol and implementation guide will be made available as well. The study coordinator will be responsible for creating these documents and maintaining them throughout the course of the study, with oversight from Dr. Rhee. External investigators interested in these materials can contact Dr. Rhee via email.
Supporting Information: Study Protocol, SAP
Time Frame: This information will be available 1 year after the publication of the first outcomes manuscript.
Access Criteria: Researchers will be able to request this information by providing a detailed analysis plan or reason for the request. They may be able to obtain de-identified individual level data with this request once the proposal has been vetted and approved. Interested parties should contact Dr. Rhee via email.

REFERENCES:
- [Background] Becan JE, Bartkowski JP, Knight DK, Wiley TRA, DiClemente R, Ducharme L, Welsh WN, Bowser D, McCollister K, Hiller M, Spaulding AC, Flynn PM, Swartzendruber A, Dickson MF, Fisher JH, Aarons GA. A model for rigorously applying the Exploration, Preparation, Implementation, Sustainment (EPIS) framework in the design and measurement of a large scale collaborative multi-site study. Health Justice. 2018 Apr 13;6(1):9. doi: 10.1186/s40352-018-0068-3. PMID 29654518
- [Background] Holtrop JS, Estabrooks PA, Gaglio B, Harden SM, Kessler RS, King DK, Kwan BM, Ory MG, Rabin BA, Shelton RC, Glasgow RE. Understanding and applying the RE-AIM framework: Clarifications and resources. J Clin Transl Sci. 2021 May 14;5(1):e126. doi: 10.1017/cts.2021.789. eCollection 2021. PMID 34367671
- [Background] McCreight MS, Rabin BA, Glasgow RE, Ayele RA, Leonard CA, Gilmartin HM, Frank JW, Hess PL, Burke RE, Battaglia CT. Using the Practical, Robust Implementation and Sustainability Model (PRISM) to qualitatively assess multilevel contextual factors to help plan, implement, evaluate, and disseminate health services programs. Transl Behav Med. 2019 Nov 25;9(6):1002-1011. doi: 10.1093/tbm/ibz085. PMID 31170296
- [Background] Feldstein AC, Glasgow RE. A practical, robust implementation and sustainability model (PRISM) for integrating research findings into practice. Jt Comm J Qual Patient Saf. 2008 Apr;34(4):228-43. doi: 10.1016/s1553-7250(08)34030-6. PMID 18468362